CLINICAL TRIAL: NCT03508622
Title: Group Telehealth Weight Management Visits for Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Brenda Manzanarez, MS, RD, Clinical Dietitian II, Children's Hospital Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-17-00509; UL1TR001855 (NIH)
Record Dates: First submitted 2018-01-06; First posted 2018-04-26 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Pilot intervention using retrospective control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): This group will receive weight management treatment via 12 online group sessions, over 6 months. They will have Bluetooth-enabled scales that will allow them to transmit their weight data to the PI in between research visits. They will answer questionnaires and have research visits at baseline, 3 months, and 6 months.
  Interventions: Behavioral: Telehealth group sessions
- Empower (Other): This retrospective control group received standard in-clinic individualized weight management with a multi-disciplinary group of providers, via 6 monthly clinic visits, over 6 months.
  Interventions: Behavioral: Empower clinic

INTERVENTIONS:
Behavioral: Telehealth group sessions — Telehealth sessions will utilize an online meeting platform and will be conducted by RDs, PTs, psychologists, and MDs, to deliver weight management information/counseling, to group of 5-6 14-18 yos with obesity.
  Arms: Telehealth
Behavioral: Empower clinic — Empower visits for the retrospective control group were multi-disciplinary in nature, occurred at CHLA outpatient clinic, and were intended to be monthly (though actual adherence to recommended attendance was variable). Teen and minimum of one family member were asked to attend monthly visits, as per our standard clinical care.
  Arms: Empower

SUMMARY:
Summary Description

The goal of this intervention study is to test how well does a weight management curriculum work in virtual group-based medical visits (telehealth) for the treatment of adolescents with obesity. The main questions it aims to answer are:

* How well does providing group-based medical care for obesity using telehealth work?
* How doable is it to provide virtual group-based health education visits with adolescent patients?
* Are the group-based health education visits similar, or better than the traditional in-person clinic visits?

Participants will be asked to:

* Complete surveys, do bloodwork, and physical measurements like blood pressure, height and weight before the study activities start and after completing the study activities
* Participate in study activities such as attending 12 virtual sessions lasting 60 minutes each, every other week, over a period of 6 months
* Join group learning and discussions of topics like nutrition, barriers to physical activity, and mental health with various facilitators like a medical doctor, dietitian, psychologist, and physical therapist
* Take part of in brief individual coaching sessions over email or over the phone Researchers will compare the virtual group-based medical visits to the traditional in-person weight management clinic visits (EMPOWER Weight Management Clinic) to see if the study can be another option in the treatment of adolescents with obesity.

DETAILED DESCRIPTION:
Background

As noted above, EMPOWER was a multi-disciplinary, team-based clinic model, involving physicians, psychologists, registered dietitians (RDs), and physical therapists (PTs) providing tertiary care management of obesity. Data from the first two years of EMPOWER showed that patients with four or more visits (n=109) experienced a decrease in average BMI z-score (-0.09SD). This, though modest, is promising; however, both cost and patient retention present significant challenges to EMPOWER and other tertiary care pediatric obesity programs, and may be barriers to further progress. Much administrative personnel time was consumed in working with insurers in order to authorize visits, and nevertheless, this type of hospital-based care was poorly reimbursed. Getting to Children's Hospital Los Angeles (CHLA) is often a major challenge for our patients, due to the large urban sprawl of Los Angeles, traffic, limited and expensive parking, and poor public transportation. Frequent visits result in missed work and school days, a burden to families. Adolescent patients face even greater challenges, as they learn to manage their own health and balance the emotional and social changes required in the transition to adulthood, with family and parental expectations and limitations.

Telehealth technology presents an innovative, cost-effective, and often highly-engaging alternative to in-person visits, which bypasses many of the logistical difficulties of getting to CHLA. Moreover, adolescents today are highly attuned to, and aligned with, digital and mobile technologies, and are natural consumers of media in this format. There is strong evidence from numerous published studies that telehealth can be an effective tool for chronic disease management. Additionally, many youth with obesity are significantly socially isolated, and our current individual patient-provider model does not effectively address this isolation in the way we expect a group session will; various published studies of group treatment have demonstrated inter-participant support and positive effects of social interaction.

While Empower's current model leads to successful weight management in many of its patients, that success is often modest, as alluded to above; and for some of patients, it simply does not work. With this study, the investigators intend to pilot a group telehealth model targeted at adolescents with obesity.

Specifically, the investigators aim to:

1. Pilot a new care delivery model for CHLA EMPOWER patients using group telehealth visits.
2. Assess the feasibility of using telehealth with adolescent patients
3. Test the efficacy of group health education sessions using video conference technology

Hypotheses:

1. Use of group health education sessions using video conference technology is a feasible, cost-effective care delivery model for adolescents being treated for obesity.
2. Efficacy of this model will be comparable to, or better than, standard multi-disciplinary in-person visits. This will be measured by:

   a. Clinical and anthropomorphic data: i. Changes in Body Mass Index (BMI), BMI percentile, and BMI percent of the 95th percentile ii. Change in blood pressure percentile iii. Change in hemoglobin A1C, ALT, triglycerides b. Quality of life c. Self-efficacy d. Satisfaction
3. Attendance to telehealth visits will be better than attendance to standard in-person visits, as measured by no-show rates and same-day reschedules

Methods and study design:

Youth 14-18 years of age who meet EMPOWER clinic criteria and consent to the study will be prospectively assigned to the intervention telehealth group (n=24); they will be compared to a restrospective cohort of "standard care" EMPOWER patients (n=24). Since the investigators do not expect a statistically significant difference in BMI change between the telehealth intervention and standard EMPOWER, power calculations were conducted on change scores in Quality of Life indicators. Using Optimal Design software v1.77 and specifying a = 0.05, anticipated effect size δ = 0.40, between-group variance ranging around 0.05, and controlling for effects of the covariates on various measures at 3 and 6 months, it is expected that 24 participants per condition will provide a moderate power to identify a treatment effect for proof of concept purposes.

The intervention group will receive:

* Group telehealth sessions twice per month for 6 months. The group sessions will be 60 minutes and involve delivery of a semi-structured curriculum including topics such as nutrition education, reducing barriers to physical activity, and mindfulness techniques. Sessions will be facilitated by EMPOWER providers (physicians, psychologists, RDs, and PTs) who will use a combination of: 1) motivational interviewing techniques, modified for the group setting, 2) supportive exploration of barriers to behavior change and 3) setting SMART goals.
* Brief individualized coaching by the program coordinator between sessions via telephone or email. It will be comparable to the personalized feedback and motivation provided in standard EMPOWER.
* Parent newsletters will be sent out monthly to inform parents of key messages; parents will also be informed of their child's attendance to the session

Control subjects received the standard EMPOWER model consisting of monthly in person clinic visits where they met individually with a combination of providers (physician, RD, PT, and/or psychologist).

The intervention group participants will have in-person visits at baseline, 3 and 6 months to measure weight, vertical growth, and blood pressure, and complete questionnaires assessing quality of life, self-efficacy and satisfaction. Anthropomorphic measures and attendance rates will be compared to the retrospective control group.

ELIGIBILITY:
Inclusion Criteria:

* Class 2 or 3 obesity OR
* Class 1 obesity plus a significant comorbidity, such as impaired glucose tolerance or type 2 diabetes mellitus, hypertension, hyperlipidemia, non-alcoholic fatty liver disease (NAFLD), polycystic ovarian syndrome (PCOS), or obstructive sleep apnea.

Exclusion Criteria:

* Significant intellectual or neurodevelopmental disability
* Inability to stand on a scale independently without assistance or use of an assistive device
* Non-English speaking

Given the shared nature of group appointments, participants should be at approximately the same developmental stage as their peers. Discussion topics may include stigma, body image, family dynamics, and school issues, and therefore a wide variance in age range or cognitive status could potentially diminish the effectiveness of the group sessions. Non-English speaking youth will be excluded due to limitations in translation services for such a small pilot project. English speaking adolescents with non-English speaking parents will be included.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Manzanarez, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Bashshur RL, Shannon GW, Smith BR, Alverson DC, Antoniotti N, Barsan WG, Bashshur N, Brown EM, Coye MJ, Doarn CR, Ferguson S, Grigsby J, Krupinski EA, Kvedar JC, Linkous J, Merrell RC, Nesbitt T, Poropatich R, Rheuban KS, Sanders JH, Watson AR, Weinstein RS, Yellowlees P. The empirical foundations of telemedicine interventions for chronic disease management. Telemed J E Health. 2014 Sep;20(9):769-800. doi: 10.1089/tmj.2014.9981. Epub 2014 Jun 26. PMID 24968105
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K, Scott RE. Home telehealth for chronic obstructive pulmonary disease: a systematic review and meta-analysis. J Telemed Telecare. 2010;16(3):120-7. doi: 10.1258/jtt.2009.090812. Epub 2010 Mar 2. PMID 20197355
- [Background] Harris MA, Freeman KA, Duke DC. Seeing Is Believing: Using Skype to Improve Diabetes Outcomes in Youth. Diabetes Care. 2015 Aug;38(8):1427-34. doi: 10.2337/dc14-2469. Epub 2015 Jun 1. PMID 26033508
- [Background] Markowitz JT, Laffel LM. Transitions in care: support group for young adults with Type 1 diabetes. Diabet Med. 2012 Apr;29(4):522-5. doi: 10.1111/j.1464-5491.2011.03537.x. PMID 22150392
- [Background] Kulik N, Ennett ST, Ward DS, Bowling JM, Fisher EB, Tate DF. Brief report: A randomized controlled trial examining peer support and behavioral weight loss treatment. J Adolesc. 2015 Oct;44:117-23. doi: 10.1016/j.adolescence.2015.07.010. Epub 2015 Aug 7. PMID 26265590
- [Background] Tanofsky-Kraff M, Shomaker LB, Young JF, Wilfley DE. Interpersonal psychotherapy for the prevention of excess weight gain and eating disorders: A brief case study. Psychotherapy (Chic). 2016 Jun;53(2):188-94. doi: 10.1037/pst0000051. PMID 27267503

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental - Telehealth: This group will receive weight management treatment via 12 online group sessions, over 6 months. They will have Bluetooth-enabled scales that will allow them to transmit their weight data to the PI in between research visits. They will answer questionnaires and have research visits at baseline, 3 months, and 6 months.
  Telehealth group sessions: Telehealth sessions will utilize an online meeting platform and will be conducted by RDs, PTs, psychologists, and MDs, to deliver weight management information/counseling, to group of 5-6 14-18 yos with obesity.
- Control - EMPOWER Clinic: This retrospective control group received standard in-clinic individualized weight management with a multi-disciplinary group of providers, via 6 monthly clinic visits, over 6 months.
  Empower clinic: Empower visits for the retrospective control group were multi-disciplinary in nature, occurred at CHLA outpatient clinic, and were intended to be monthly (though actual adherence to recommended attendance was variable). Teen and minimum of one family member were asked to attend monthly visits, as per our standard clinical care.
Period: Overall Study
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Started | 33 | 33
Completed | 15 | 9
Not Completed | 18 | 24
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 16 | 0
Not completed — Incomplete data | 0 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 8
  Between 18 and 65 years | 26 | 30 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.27 (1.52) | 15.51 (3.84) | 15.88 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 12 | 15 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 0 | 0
  Race: Asian or Pacific Islander | 1 | 0 | 1
  Race: Black/African American | 1 | 0 | 1
  Race: Hispanic/Latino | 13 | 3 | 16
  Race: White/Caucasian | 2 | 9 | 11
  Race: Unknown | 9 | 6 | 15
  Race: Other | 4 | 15 | 19
  Race: Non-Hispanic | 0 | 0 | 0
  Race: Mexican | 1 | 0 | 1
  Ethnicity: American Indian or Alaskan Native | 1 | 0 | 1
  Ethnicity: Asian or Pacific Islander | 0 | 0 | 0
  Ethnicity: Black/African American | 3 | 0 | 3
  Ethnicity: Hispanic/Latino | 26 | 20 | 46
  Ethnicity: White/Caucasian | 1 | 0 | 1
  Ethnicity: Unknown | 0 | 6 | 6
  Ethnicity: Other | 0 | 1 | 1
  Ethnicity: Non-Hispanic | 0 | 6 | 6
  Ethnicity: Mexican | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 6 Months in Body Mass Index
Description: A measure for body adiposity calculated by dividing a participant's weight in kilograms by the square of their height in meters (kg/m^2)
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: kilograms by the square of their height
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 31 | 33
kilograms by the square of their height | 1.07 (2.06) | 0.17 (1.43)

2. Primary Outcome: Mean Change From Baseline to 6 Months in Percentage of 95th Percentile Body Mass Index
Description: A measure of body adiposity for severe obesity calculated by dividing a participant's weight in kilograms by the square of their height in meters (kg/m^2) and categorized as per the American Academy of Pediatrics
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: percent 95th percentile body mass index
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 31 | 33
percent 95th percentile body mass index | 1.62 (6.84) | -2.52 (4.66)

3. Primary Outcome: Mean Change From Baseline to 6 Months in Glycosylated Hemoglobin
Description: a blood test that measures the average blood glucose over three months
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 31 | 33
mg/dL | -0.27 (.85) | -.16 (0.24)

4. Primary Outcome: Mean Change From Baseline to 6 Months in Alanine Aminotransferase
Description: Alanine Aminotransferase (ALT) will be assessed via blood test measured in units/liter. The range from 7 to 56 units per liter (U/L) of blood indicates normal levels and, 57 and greater indicate elevated levels.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 15 | 9
units per liter (U/L) | 18.8 (156.00) | 3.00 (24.6)

5. Primary Outcome: Mean Change in Triglycerides From Baseline to 6 Months
Description: Triglycerides will be assessed via blood tests and measured in milligrams per deciliter (mg/dL).
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 31 | 33
milligrams per deciliter (mg/dL) | -7.2 (70.31) | -44.71 (124.13)

6. Primary Outcome: Mean Change in Diastolic Blood Pressure From Baseline to 6 Months
Description: Blood pressure will be assessed via a blood pressure monitor (a device used to measure blood pressure) measured in millimeters of mercury (mmHg). Systolic mmHg less than 70 indicates normal level, above 70 indicates elevated level, and Diastolic mmHg less than 120 indicates normal level, and above 120 indicates elevated level.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 15 | 33
millimeters of mercury (mmHg) | -2.47 (6.8) | -2.88 (9.81)

7. Primary Outcome: Mean Change in Systolic Blood Pressure From Baseline to 6 Months
Description: as for outcome 6
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 15 | 33
millimeters of mercury (mmHg) | 4.1 (10.1) | -4.82 (9.74)

8. Secondary Outcome: Change in Quality of Life From Baseline to 6 Months Using Quality of Life Questionnaire #1
Description: Quality of life measurements will be obtained will be obtained through "Youth Telehealth Pilot Study Survey" questionnaire. Questionnaire with a scale from 1 (only a little), 3 (some) to 5 (a lot). Mean will be provided to describe change.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental - Telehealth
Number analyzed (Participants) | 17
score on a scale
  treated the same as everyone else? | 0.7 (0.7)
  accepted just as you are? | 0 (1)
  challenged and encouraged through sports? | 0.4 (1.3)
  successful or skilled in some sport or other activity you like? | 0.7 (0.6)
  happy with yourself? | 0 (0.7)
  able to speak up for yourself? | 0.9 (1.1)
  satisfied with your school day? | 0.1 (1.1)
  able to take part in group activities? | 1.0 (1.6)
  able to have a special friend? | 0.4 (1.4)
  are as independent as you are able to be? | 0.1 (0.9)
  have the physical strength to do sports like swimming, soccer, basketball, etc? | 0.5 (0.9)
  How much do you feel that you: have a lot of pain? | -0.4 (0.9)
  How much do you feel that you: can speak up for yourself? | 0.2 (1.4)
  How much do you feel that you can make your own choices and decisions? | -.05 (0.8)
  How much do you feel that you: are treated the same as the other kids? | 0.2 (0.8)
  How much do you feel that you: are positive about yourself? | 0.1 (0.7)
  How much do you feel that: other people respect you? (not teased; include you in activities) | 0.05 (0.8)
  you have a say in your medical treatment? | 0.2 (1.35)
  How much do you feel that: you understand the long term health impacts of being overweight? | -0.1 (0.7)
  How much do you feel that: people see you for who you are? | 0.2 (0.8)
  How much do you feel that: you are able use the kitchen at home? | -0.05 (0.8)
  How much do you feel that: you participate in outdoor activities? | 0.5 (1.1)
  How much do you feel that : there is hope for the future? | 0 (0.5)
  How much do you feel that : you will have a suitable home in the future? | 0 (0.5)
  How much do you feel that : you are able to go out on dates and to parties? | 0.5 (1.1)
  How much do you feel that : there will be job opportunities for you in the future? | 0.2 (1.0)
  How much do you feel that : you are able to get an education for a job that interests you? | 0.1 (1.1)
  How much do you feel that : you have a career goal in mind? | 0.1 (0.8)
  How much do you feel that : you will be able to hold down a part-time job? | 0.5 (1.0)
  How much do you feel that : you will be able to have children in the future? | 0.4 (1.4)
  How much do you feel that : you will marry? | -0.2 (1.2)
  How much do you feel that : you have a close friend who is like you in many ways? | 0.1 (1.3)

9. Secondary Outcome: Change in Quality of Life From Baseline to 6 Months Using the Quality of Life 2 (KINDL) Questionnaire.
Description: Quality of Life measurements will be obtained through will be obtained through "Youth Telehealth Pilot Study Survey" questionnaire. Questions 1-13 on questionnaire use a scale from 1 to 5 with 1) Never, 2) Rarely, 3) Sometimes, 4) Often, 5) All the time. Question 14 uses scale from 1 to 5 with 1) Not at all, 2) Somewhat severe , 3) Moderately severe , 4) Fairly, 5) Very Severe. Question 15 on questionnaire use a scale from 1 to 5 with 1) not at all 2) Somewhat 3) Moderately, 4)A lot, 5) Really a lot
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control - EMPOWER Clinic
Number analyzed (Participants) | 31
units on a scale
  During the past week I felt so big that it was hard to move. | 0.06 (0.42)
  I got tired and out of breath quickly compared to others when being physically active. | -0.12 (0.76)
  During the past week I was sad and depressed because of my weight | -0.12 (0.90)
  During the past week I was annoyed by my many attempts at losing weight | -0.88 (1.08)
  During the past week I felt ashamed because of my weight | -.35 (0.97)
  During the past week was dissatisfied with myself because of my weight | -0.59 (1.19)
  During the past week my family scolded me because of my weight | -0.47 (1.72)
  During the past week had to eat at home because I'm watching my weight | 0.12 (1.32)
  During the past week was teased by others because of my weight | 0.12 (1.32)
  During the past week was left out by others when they did things together, because of my weight | 0.06 (1.06)
  During the past week was distracted during school by the thought of food | -0.35 (1.23)
  During the past week I was not able to take part in sports at school because of my weight | -0.29 (1.18)
  How often during the past week did you feel physically uncomfortable because of being obese? | 0.12 (0.96)
  How severe was your discomfort because of being overweight during the past week? | -0.35 (0.97)
  How much did it bother you being overweight during the past week? | -0.29 (0.96)

10. Secondary Outcome: Satisfaction With Care at 6 Months Using Satisfaction Telehealth Questionnaire
Description: Satisfaction measurements will be obtained through "Satisfaction using Telehealth" questionnaire.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental - Telehealth
Number analyzed (Participants) | 17
Participants
  I felt comfortable using technology for my online sessions.: Agree or Strongly Agree | 13
  I felt comfortable using technology for my online sessions.: Neutral | 4
  I felt comfortable using technology for my online sessions.: Disagree or Strongly Disagree | 0
  Participating in the TH sessions was much easier than going in person doctor's appointment.: Agree or Strongly Agree | 10
  Participating in the TH sessions was much easier than going in person doctor's appointment.: Neutral | 7
  Participating in the TH sessions was much easier than going in person doctor's appointment.: Disagree or Strongly Disagree | 0
  I would like to have online sessions again.: Agree or Strongly Agree | 8
  I would like to have online sessions again.: Neutral | 9
  I would like to have online sessions again.: Disagree or Strongly Disagree | 0
  I liked talking to other teens and young adults during the online sessions.: Agree or Strongly Agree | 5
  I liked talking to other teens and young adults during the online sessions.: Neutral | 12
  I liked talking to other teens and young adults during the online sessions.: Disagree or Strongly Disagree | 0
  I felt supported during the group sessions.: Agree or Strongly Agree | 14
  I felt supported during the group sessions.: Neutral | 3
  I felt supported during the group sessions.: Disagree or Strongly Disagree | 0
  I felt comfortable asking the session leader questions throughout the online sessions.: Agree or Strongly Agree | 12
  I felt comfortable asking the session leader questions throughout the online sessions.: Neutral | 5
  I felt comfortable asking the session leader questions throughout the online sessions.: Disagree or Strongly Disagree | 0
  I was able to speak freely and express myself.: Agree or Strongly Agree | 14
  I was able to speak freely and express myself.: Neutral | 3
  I was able to speak freely and express myself.: Disagree or Strongly Disagree | 0
  I felt comfortable showing my face with others on screen during the sessions.: Agree or Strongly Agree | 3
  I felt comfortable showing my face with others on screen during the sessions.: Neutral | 9
  I felt comfortable showing my face with others on screen during the sessions.: Disagree or Strongly Disagree | 5
  I liked the group style of the sessions.: Agree or Strongly Agree | 10
  I liked the group style of the sessions.: Neutral | 7
  I liked the group style of the sessions.: Disagree or Strongly Disagree | 0
  I felt that the check-ins between sessions helped me stay motivated to work on my goals/activities.: Agree or Strongly Agree | 9
  I felt that the check-ins between sessions helped me stay motivated to work on my goals/activities.: Neutral | 6
  I felt that the check-ins between sessions helped me stay motivated to work on my goals/activities.: Disagree or Strongly Disagree | 2
  I felt that the check-ins helped me to follow through with my goals and photovoice activities.: Agree or Strongly Agree | 12
  I felt that the check-ins helped me to follow through with my goals and photovoice activities.: Neutral | 5
  I felt that the check-ins helped me to follow through with my goals and photovoice activities.: Disagree or Strongly Disagree | 0
  I would recommend telehealth as a form of receiving personalized health care and medical information: Agree or Strongly Agree | 12
  I would recommend telehealth as a form of receiving personalized health care and medical information: Neutral | 5
  I would recommend telehealth as a form of receiving personalized health care and medical information: Disagree or Strongly Disagree | 0
  I enjoyed watching the videos that were shown and discussed during the online sessions.: Agree or Strongly Agree | 13
  I enjoyed watching the videos that were shown and discussed during the online sessions.: Neutral | 4
  I enjoyed watching the videos that were shown and discussed during the online sessions.: Disagree or Strongly Disagree | 0
  I am satisfied with the health care and medical information that I received for weight management: Agree or Strongly Agree | 15
  I am satisfied with the health care and medical information that I received for weight management: Neutral | 2
  I am satisfied with the health care and medical information that I received for weight management: Disagree or Strongly Disagree | 0
  The session leader provided education that was easy to understand: Agree or Strongly Agree | 15
  The session leader provided education that was easy to understand: Neutral | 2
  The session leader provided education that was easy to understand: Disagree or Strongly Disagree | 0

11. Secondary Outcome: Attendance/Retention From Baseline to 6 Months
Description: Attendance, no-show and same-day reschedules
Time Frame: Baseline to 6 Months
Measure: Mean (Inter-Quartile Range); unit: patient visits
Arm/Group | Experimental - Telehealth | Control - EMPOWER Clinic
Number analyzed (Participants) | 16 | 33
patient visits | 6.9 [1 to 12] | 5.5 [5 to 7]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Telehealth | Empower
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

LIMITATIONS AND CAVEATS:
This study is limited by a relatively small sample size (intervention n = 31, control n=33) and short duration of follow-up (6 months). Study did not reach target number to achieve target power and statistical reliability. Therefore, results should be interpreted with caution until a larger scale and more rigorous study is replicated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03508622/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03508622/ICF_001.pdf